CLINICAL TRIAL: NCT04831307
Title: Evaluation of the in Vivo Biodistribution and Radiation Dosimetry of 68Ga-HTK03149 for Use as a Diagnostic Radiopharmaceutical
Brief Title: 68Ga-HTK03149 for Use as a Diagnostic Radiopharmaceutical
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H21-00749
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer; Prostatic Neoplasm; Prostatic Disease; Urogenital Neoplasms; Disease Attributes; Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Urogenital Neoplasms; Disease Attributes; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-HTK03149 PET/CT (Experimental): 200 MBq/m2 of body surface area, with a 200 MBq minimum adult administered activity will be injected intravenously prior to perform the PET/CT
  Interventions: Other: [68Ga]Ga-HTK03149 PET/CT

INTERVENTIONS:
Other: [68Ga]Ga-HTK03149 PET/CT — 200 MBq/m2 of body surface area, with a 200 MBq minimum adult administered activity will be injected intravenously prior to perform the PET/CT

SUMMARY:
This is a preliminary evaluation of a radiotracer's biodistribution in human subjects. It is a prospective, single-centre, open-label, single group assignment interventional study.

Prostate cancer is very common, and PSMA imaging is currently the most accurate means of localizing these tumours.

The goal is to evaluate the biodistribution and safety of [68Ga]HTK03149 PET/CT for prostate cancer imaging.

DETAILED DESCRIPTION:
Each subject will have a PET/CT scan using [68Ga]HTK03149 . The [68Ga]HTK03149 radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada.

After providing informed written consent subjects will complete a medical history questionnaire.

Monitoring of adverse events There will be short-term evaluation of adverse events by comparison of vital signs before and after administration of [68Ga]HTK03149 . Eighteen to seventy-two hours after [68Ga]HTK03149 administration the participant will return to the imaging department to perform a follow up safety assessment and routine blood draw. The study coordinator will ask the participant if they have experienced any adverse events during that time period and complete the adverse event questionnaire.

Follow-up Assessments

The following information will be collected up to 12 months following the PET/CT scans:

Initiation of a new treatment, Laboratory results and pathology reports, Results of imaging studies, Final clinical diagnosis by physician and relevant clinical notes. The study is expected to take up to 1 year for accrual.

ELIGIBILITY:
Inclusion Criteria:

* Participants with newly diagnosed or documented prostate cancers (PCa), with at least one measurable lesion based on CT, MR or at least one visualised lesion on PET/CT imaging (either from an 18F-DCFPyL or 68Ga-PSMA-11 PET).
* ECOG performance status of 2 or less.

Exclusion Criteria:

* Medically unstable (eg. acute illness, unstable vital signs)
* Unable to lie supine for the duration of imaging
* Unable to provide written consent
* Exceeds safe weight limit of the PET/CT bed (204.5 kg) or unable to fit through the PET/CT bore (diameter 70 cm)
* Patients with widespread liver metastases occupying more than 50% of the liver volume will not be eligible to participate in this study as this would preclude assessment of normal liver activity for dosimetry purposes.
* Patients with baseline ALT or AST higher than 5× ULN or 250 U/L.
* Patients with elevated baseline levels of total bilirubin (higher than 1.2× ULN, or 1.3 mg/dL, (with exception of Gilbert's syndrome), with INR >1.2, or platelet count below the lower limit of normal (typically <150 000/μL.
* Patients with elevated alkaline phosphatase (ALP), equal to or higher than 2× ULN or 250 U/L, unless the ALP elevation is not from a hepatic origin.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of 68Ga-HTK03149 PET/CT in human subjects | Up to 12 months
  Evaluate the biodistribution of 68Ga-HTK03149 in human subjects, which will enable calculating the radiation dosimetry of this radiopharmaceutical. The efficacy parameters will be the following:
  Individual organ dose and effective dose measured in mSV/MBq. Descriptive statistics on normal organ and tumour uptake reported in standardized uptake values (SUV).
  Tumour/blood, tumour/liver, tumour/kidney and tumour/lung ratios will be reported.

SECONDARY OUTCOMES:
Number of participants with 68Ga-HTK03149 related adverse events as assessed by abnormal vital sign measurement | Before injection, 1 hours post injection, 2 hours post injection and 2.5 hours post injection
  Vital signs (blood pressure, heart rate and pulse oximetry) will be measured at four time points. All values that fall outside of the normal parameters will be assessed by a physician and reported as an adverse event.
Number of participants with self-reported 68Ga-HTK03149 related adverse event | 18-72 hours
  Patients will return to the department 18-72 hours after the 68Ga-HTK03149 PET/CT scan to see if they experienced any adverse events. These are recorded and evaluated for severity and likelihood they are related to the study drug. All adverse events will be recorded and summarized in the final report.
Perform a preliminary assessment of 68Ga-HTK03149 uptake in prostate cancer lesions | Up to 12 months
  Determination of tumour uptake will be performed by contouring the tumours using a threshold to match the size of the lesion on CT imaging. The standardized uptake value (SUV) will be calculated and normalized for both body weight and lean body mass (SUVlean). The maximal, mean and peak (activity in the highest 1 cc voxel cluster) will be determined and recorded. The tumour/blood, tumour/liver and tumour/lung ratios will be reported for descriptive analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada